CLINICAL TRIAL: NCT00485602
Title: Orthodontic Treatment With a Part-Time Wearing Esthetic Removable Appliance
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAFENALIGN-HMO-CTIL
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Malocclusion
Keywords: malocclusion; aligner; crowding; expansion; orthodontic treatment
MeSH Terms: conditions — Malocclusion; Crowding | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: orthodontic treatment with "Rafenalign" appliance

SUMMARY:
The trial is aimed to investigate an orthodontic treatment with a new removable-part-time-wearing appliance, based on "High-Tech" technology.

The appliance should be wear only 12-14 hours a day, and is made of a single silicone aligner, made specifically for the patient, using 3-D screening technology of the patient's malocclusion. The aligner has a designed pathway "built-in" for the tooth to move, from the original position of the malocclusion to the "end point" - the correct position.

The force system, that is needed in order to generate tooth movement, is produced by tiny air-balloons which are incorporated in the aligner.

The study hypothesis is, that an orthodontic treatment can be done successfully with this part-time wearing appliance.

DETAILED DESCRIPTION:
The appliance include:

* silicone aligner (made specifically for the patient.
* simple air pump to blow air in the tiny balloons.

The patient is guided to wear the appliance 12-14 hours a day, after filling air in the balloons, under the doctor's instructions.

Clinical examination for follow-up will be done every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate class I malocclusion
* good general health
* good oral hygiene

Exclusion Criteria:

* bad cooperation
* any mental or health problem
* severe class I malocclusion, class II or class III malocclusion

Ages: 8 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
study models | every 2 appointments (8 weeks)

SECONDARY OUTCOMES:
occlusal photographs | every 3 appointments (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Redlich, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel